CLINICAL TRIAL: NCT01875172
Title: Smoking Cessation in Pregnancy: A Pilot Study Comparing Counseling With and Without Sustained-Release Bupropion
Brief Title: Bupropion for Smoking Cessation in Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watching Over Mothers & Babies Foundation (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Hugh Miller, Medical Director, Watching Over Mothers & Babies Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21CA089510-01A2 (NIH)
Record Dates: First submitted 2013-04-14; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Smoking Cessation; Pregnancy
Keywords: bupropion SR; randomized controlled trial; pregnancy
MeSH Terms: conditions — Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion SR (Experimental): Study medication (150 mg bupropion SR) daily for 14 days. Women still smoking at 2-weeks & 4-weeks were encouraged to increase their medication to two times per day (150 mg bid). Women received smoking cessation counseling at baseline, 2, 4, 6, and 8 weeks.
  Interventions: Drug: Bupropion SR; Behavioral: smoking cessation counseling
- Placebo (Placebo Comparator): Study medication (placebo) daily for 14 days. Women still smoking at 2-weeks & 4-weeks were encouraged to increase their medication to two times per day. Women received smoking cessation counseling at baseline, 2, 4, 6, and 8 weeks.
  Interventions: Drug: placebo; Behavioral: smoking cessation counseling

INTERVENTIONS:
Drug: Bupropion SR — Comparison of bupropion SR or placebo + smoking cessation counseling
  Other Names: Wellbutrin SR; Zyban SR
  Arms: Bupropion SR
Drug: placebo
  Arms: Placebo
Behavioral: smoking cessation counseling

SUMMARY:
The purpose of this study is to determine whether bupropion SR increases cessation and/or smoking reduction among pregnant smokers.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of a pharmacologic agent (bupropion SR) to achieve higher rates of smoking cessation and greater reduction in smoking during pregnancy

Secondary Objective:

To evaluate the safety of using a pharmacologic agent (bupropion SR) for smoking cessation in pregnancy.

Hypotheses to be tested:

1. Bupropion SR combined with smoking cessation counseling during pregnancy will increase smoking cessation, compared to smoking cessation counseling combined with placebo, or standard of care.
2. Bupropion SR combined with smoking cessation counseling during pregnancy will produce greater reduction in smoking in patients unable to quit, as compared to smoking cessation counseling combined with placebo, or standard of care.
3. Bupropion SR combined with smoking cessation counseling during pregnancy will improve perinatal outcomes (by decreasing preterm birth, preterm premature rupture of membranes, antenatal bleeding, low birth weight, intrauterine growth restriction and increasing maternal weight gain), as compared to smoking cessation counseling combined with placebo, or standard of care.
4. Bupropion SR combined with smoking cessation counseling during pregnancy will increase the rate of smoking cessation without increasing the number of adverse events reported by women, as compared to smoking cessation counseling combined with placebo, or standard of care.

Few studies have offered pregnant women pharmacologic assistance with their tobacco addiction for the purpose of achieving smoking cessation in pregnancy. In view of the evidence from the non-pregnant population, pharmacologic assistance with either nicotine replacement therapy or bupropion is essential to significant cessation and reduction programs. This pilot study is designed to generate sufficient preliminary data to support future grant applications to state and/or federal funding agencies for adequate funding to conduct a properly powered randomized clinical trial. This pilot study will provide useful information for future sample size calculations and give some indication as to the rate of adverse reactions and safety profile of bupropion taken during pregnancy.

Cigarette smoking is associated with various complications of pregnancy., Likewise, infants and children of women who smoke during pregnancy are at greater risk for a myriad of physical and developmental problems. Women who participate in the study and receive the intervention may benefit if they reduce or stop their tobacco use. Decreased cigarette smoking by pregnant subjects enrolled in this study may lead to a reduction in complications of pregnancy and health problems of infants and children that are attributable to smoking.

The standard therapy for pregnant women is to receive some directive counseling from their clinician. Occasionally, patients will even be referred to community organizations to reinforce the office counseling. The evidence suggests that there is limited value to behavioral counseling alone and that most clinicians are not properly trained and that those who are, do not have the time to adequately counsel patients. There are no smoking cessation programs currently available in the Tucson community that offer pharmacologic assistance in combination with counseling to pregnant women. Individual clinicians do prescribe pharmacologic aids for their patients on a case by case basis.

Smoking cessation counseling is evidence based. However, as the investigators have previously indicated it is rarely conveyed to patients because of inadequate training and time. There is currently no support within obstetrical healthcare funding to subsidize the cost of this service.

ELIGIBILITY:
Inclusion Criteria:

* Smoked at least one puff in the past 7 days
* Confirmed viable gestation

Exclusion Criteria:

* All patients found to have a non-viable fetus or major congenital anomaly
* History of seizure disorder
* Family history of seizure disorder
* History of severe head trauma
* History of anorexia nervosa or bulimia
* Current use of nicotine-replacement therapy
* Unstable medical or psychiatric condition
* Current use of an monoamine oxidase inhibitor or bupropion hydrochloride products

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2001-10; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
biologically verified smoking cessation or reduction | 8 weeks and delivery
  change in smoking from study enrollment to end of treatment (8 weeks) and at delivery

SECONDARY OUTCOMES:
adverse events reported during pregnancy | 8 weeks and delivery
self reported smoking cessation or reduction | 8 weeks and delivery
  change in self reported smoking from study enrollment to end of treatment (8 weeks) and at delivery

OTHER OUTCOMES:
depression | 8 weeks and delivery
  change in depression (measured by the Edinburgh postnatal depression scale) between study enrollment and end of treatment (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh S Miller, MD, Principal Investigator — Watching Over Mothers and Babies Foundation
Locations (1):
- Watching over Mothers and Babies Foundation, Tucson, Arizona, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961